CLINICAL TRIAL: NCT06659276
Title: Whole Body DWI Sequences As Compared with Standard FDG PET/CT in Patients with Simptomatic Multiple Myeloma
Brief Title: Comparison Between Whole Body DWI and FDG PET/CT in Patients with Simptomatic Multiple Myeloma
Acronym: MMR-PET-22-04
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Cristina Nanni, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: IRCCS S.Orsola Malpighi
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma, staging, therapy assessment, DWI, FDG PET CT
MeSH Terms: conditions — Multiple Myeloma; Driving Under the Influence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with new diagnosis of symptomatic multiple myeloma: fdg pet/CT and Whole body MRI with DWI

SUMMARY:
The primary objective is to evaluate the concordance of FDG PET/CT and total body DWI MRI sequences performed during staging and at the completion of therapy. Specifically, we will assess the positivity rates, both patient-based and lesion-based (total and by district), of the two methods during staging and at the completion of therapy. An interim analysis will be conducted comparing the two methods, followed by a final prognostic analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with symptomatic myeloma in the staging phase or with suspected symptomatic myeloma in the diagnostic phase

  * Patients who have signed the informed consent form

Exclusion Criteria:

* Patients simultaneously affected by other neoplastic diseases or with a history of other neoplasms in the previous 5 years

  * Age < 18 years
  * Women who are breastfeeding or pregnant
  * Patients with metal implants or devices that constitute an absolute contraindication for MRI
  * Patients with severe claustrophobia
  * Patients with bone pain that prevents prolonged maintenance of the supine position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: no additional info
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
positivity rate | 33 months
  comparison per patient and per lesion between FDG PET CT and WB DWI

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico S.Orsola Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided